CLINICAL TRIAL: NCT06562517
Title: Development of a Digital Training Module for Sustainable Education of Pediatric Oncology Nurses and Evaluation of Its Effectiveness
Brief Title: Digital Training Module for Sustainable Education of Pediatric Oncology Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Teaching and Research Assistant, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KOCUNI
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Cancer
Keywords: education; nursing; development; pediatric oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled pre-test-post-test design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-Standard care (No Intervention): No intervention will be performed on the nurses in this group. After the research is completed, access to the website will be provided to the nurses in the control group.
- Intervention Group (Experimental): The group will use the digital training modules developed for sustainable pediatric oncology nursing education for six months.
  Interventions: Other: Digital training module

INTERVENTIONS:
Other: Digital training module — The intervention is a 24/7 accessible educational website for pediatric oncology nurses, based on the EONS Cancer Nursing Education Framework. It features five validated training modules, enhanced with visual and auditory materials such as videos and infographics. Nurses will receive login credentials, allowing them to access the platform and participate in the training. Each module ends with a 20-question test, requiring a score of 60 to advance. A support line enables nurses to ask questions directly to researchers. Successful completion of each module earns a certificate. The website will be piloted with 15 nurses, and feedback will be used to refine its design and content.
  Arms: Intervention Group

SUMMARY:
Pediatric oncology nurses are healthcare professionals who constantly communicate with children and their families for 24 hours, and take professional roles and responsibilities in areas such as care planning, a continuation of treatment, and symptom management.However, there is no standard undergraduate education program accepted worldwide in the field of pediatric oncology nursing. For example, undergraduate nursing education in Türkiye is carried out in line with the Nursing National Core Education Program (NNCEP), and information about pediatric oncology nursing is included in the curriculum of specific courses in undergraduate programs. In addition, nurses graduate without specializing in any field in our country. Therefore, the education of pediatric oncology nurses and the continuity of education is an essential problem in developing and low-middle-income countries like our country. This prospective study in randomized controlled pre-test-post-test design aimed to develop an online website consisting of information and support modules for the care of children with cancer for sustainable pediatric oncology nursing education in Türkiye.

DETAILED DESCRIPTION:
In developed countries, there are various programs for pediatric oncology nurses to improve the quality of nursing care. Unfortunately, the inadequacy of these education programs in developing countries may prevent childhood cancer patients from receiving advanced care but may cause health inequalities. For this reason, it is very important to strengthen pediatric oncology nurses in terms of education and to develop platforms that will provide education continuity in low and middle-income countries. Today, one of the methods used to ensure the continuity and easy accessibility of education is digital education programs. Web-based education programs can increase nurses' knowledge and competence in related care issues. In studies, nurses state that planned educations were beneficial and increased their knowledge level. An accessible and sustainable web-based standard education program will enable nurses to become more competent in pediatric oncology and increase the quality of care. In Türkiye, which is a middle-income country, there is no standard curriculum for pediatric oncology nurses. Although pediatric oncology nursing is partially included in the oncology nursing certification program by the Oncology Nursing Association, we could say that it is insufficient to meet nurses' sustainability and educational needs. Therefore, there is a need for a digital website consisting of information and support modules to care for children with cancers for sustainable pediatric oncology nursing education in Türkiye.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Working in a pediatric oncology clinic,
* Having at least one year of experience in pediatric oncology.

Exclusion Criteria:

* Lack of Internet literacy,
* Incomplete filling of data collection forms.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric Oncology Nurses' Educational Needs Scale | It will be applied to nurses in the experimental and control groups before (1 week before) and after (immediately after and 6 months later) the intervention.
  The scale consists of five sub-dimensions: disease, chemotherapy, and its side effects, other treatments and their side effects, palliative care, and supportive care. From the scale, a minimum of 42 points and a maximum of 210 points can be obtained. The increase in the total score of the scale and the mean score of the sub-dimensions indicate that the education needs of the nurses regarding that sub-dimension have increased.
Knowledge Levels of Pediatric Oncology Nurses on Childhood Cancers and Care | It will be applied to nurses in the experimental and control groups before (1 week before) and after (immediately after and 6 months later) the intervention.
  To evaluate the knowledge levels of pediatric oncology nurses on childhood cancers and care, test questions will be created by the digital education modules.
Ateşman Readability Index | The data collection process will begin one day after the digital booklet is created.
  To determine the readability level of the digital training booklet, the Ateşman Readability Index will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Eyşan Hanzade Savaş, PhD, Study Chair — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No